CLINICAL TRIAL: NCT03988309
Title: Use of a Multiplexed Molecular Biomarker Test Cxbladder, in Real World Decision Making to Provide Clinical Utility Using a Randomized Design ("STRATA Study")
Brief Title: STRATA: Safe Testing of Risk for AsymptomaTic MicrohematuriA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pacific Edge Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CXB/2019/US
Record Dates: First submitted 2019-04-24; First posted 2019-06-17 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Hematuria; Urothelial Carcinoma
MeSH Terms: conditions — Hematuria; Carcinoma, Transitional Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test, subjects categorised as "low risk" or "Not low risk" (Active Comparator): A clinical risk factor nomogram risk classification will be used in this study. The nomogram categorizes subjects as either "low risk" or "not low risk" categories. "Low risk" subjects satisfy all conditions and "not low risk" satisfies at least one of the conditions.The Cxbladder Triage test result will be provided to physicians for all "low risk" subjects on the test arm. If a "low risk" subject has a Cxbladder Triage negative test result then the indication is to rule out the subject without further assessment. The decision to rule-out or further evaluate is solely that of the physician and subject. If the "low risk" subjects are not Cxbladder Triage negative then a Cxbladder Detect test result will also be provided. The indication is further evaluation as per standard of care. Subjects categorised as "not low risk" will be evaluated as per standard of care. Note that Cxbladder test results will be available for eventual analysis for these subjects.
  Interventions: Diagnostic Test: Cxbladder
- Control (No Intervention): Subjects on the control arm will be on standard of care. Trial nomogram clinical risk factor categorization for control arm subjects will not be provided to the physician (but appropriate information will be collected on the CRF to enable sub-group analysis) No Cxbladder test results will be provided for control arm subjects. Note that Cxbladder test results will be available for eventual analysis for these subjects.

INTERVENTIONS:
Diagnostic Test: Cxbladder — The Cxbladder Triage test result will be provided to physicians for all "low risk" subjects on the test arm. If a "low risk" subject has a Cxbladder Triage negative test result then the indication is to rule out the subject without further assessment. The decision to rule-out or further evaluate is solely that of the physician and subject. If the "low risk" subjects are not Cxbladder Triage negative then a Cxbladder Detect test result will also be provided. The indication is further evaluation as per standard of care. "Not low risk" patients will be evaluated as per standard of care.
  Arms: Test, subjects categorised as "low risk" or "Not low risk"

SUMMARY:
To evaluate the clinical utility associated with the integration of Cxbladder into the evaluation of subjects presenting with hematuria for evaluation of urothelial carcinoma (UC) without compromising detection of UC.

DETAILED DESCRIPTION:
Randomised two arm pragmatic clinical study to be conducted at multiple sites in US and Canada. The trial will recruit hematuria subjects, presenting to qualified sites (academic, community), who are being evaluated for urothelial carcinoma (UC). Up to 100 consecutive eligible subjects will be recruited per site.

ELIGIBILITY:
Inclusion Criteria:

* Patient is undergoing investigation of recent confirmed hematuria, as defined by the AUA/SUFU Guideline (Barocas DA, Boorjian SA, Alvarez RD et al. Microhematuria: AUA/SUFU guideline, J Urol 2020; 204:778) (by either flexible or rigid cystoscopy/TURBT), including hematuria subjects referred due to suspicious/positive imaging, in order to determine the presence of urothelial carcinoma.
* Able to provide a voided urine sample of the required minimum volume
* Able to give written consent
* Able and willing to comply with study requirements
* Aged 18 years or older

Exclusion Criteria

* Prior history of bladder malignancy or pelvic radiotherapy. Prior history prostate or renal cell carcinoma within the last 5 years.
* Prior genitourinary manipulation (flexible or rigid cystoscopy / catheterisation, urethral dilation) in the 14 days before urine collection,
* Known current pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 554 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
To measure the change in cystoscopy procedure use count between control and test arms when Cxbladder Triage is used in the evaluation | The outcome measure will be assessed by 6 months after trial completion.
  To evaluate the increase in utility as defined by the reduction in cystoscopy procedure count when Cxbladder is used in the evaluation. The comparison will be made when comparing test and control arms on a per subject basis. The gold standard for determination of a confirmed clinical diagnosis is cystoscopy confirmed by pathology, plus imaging or any follow-up investigations relating to the visit.

SECONDARY OUTCOMES:
To measure the change in total procedure use (and the invasive procedure sub-group) count between control and test arms when Cxbladder is used in the evaluation. | The outcome measure will be assessed by 6 months after trial completion.
  To evaluate the increase in utility as defined by the reduction in total procedures (and the invasive procedures subgroup) count when Cxbladder is used in the evaluation. The comparison will be made when comparing test and control arms on a per subject basis.
To measure the number of subjects who were incorrectly diagnosed associated with the integration of Cxbladder into the evaluation of subjects (or sub-cohorts on test and control arms) presenting with hematuria for evaluation of UC | The outcome measure will be assessed by 6 months after trial completion.
  To quantify the false negative rate (the percentage of the negative fraction incorrectly diagnosed) associated with the integration of Cxbladder into the evaluation of subjects (or sub-cohorts on test and control arms) presenting with hematuria for evaluation of UC
To clinically validate the performance characteristics and test negative rate of the Cxbladder Detect+ test. | The outcome measure will be assessed by 6 months after trial completion.
  The Cxbladder Detect+ test results will be compared to that of cystoscopy, which is the gold standard method for diagnosing urothelial cancer; the true positive and true negative rates will be measured, along with the false positive and false negative rates of the test. The results will be reported as sensitivity, specificity, positive and negative predictive value and test negative rate of the Cxbladder Detect+ test for detecting urothelial cancer in patients referred for evaluation of hematuria.
Quantify performance characteristics of Cxbladder signatures including for the detection of high grade/stage UC. | The outcome measure will be assessed by 6 months after trial completion.
  The Cxbladder signature test results will be compared to that of cystoscopy, which is the gold standard method for diagnosing urothelial cancer; the true positive and true negative rates will be measured, along with the false positive and false negative rates of the test. The results will be reported as sensitivity, specificity, positive and negative predictive value of the Cxbladder signature tests for detecting urothelial cancer in patients referred for evaluation of hematuria.

CONTACTS AND LOCATIONS:
Overall Officials: Tony Lough, PhD, Study Chair — Pacific Edge Pty Ltd
Locations (12):
- United States (10):
  - Institute of Urology, USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Avant Concierge Urology, Winter Garden, Florida
  - Accellacare, Chicago, Illinois
  - Allina Health Cancer Institute, Minneapolis, Minnesota
  - University of Minnesota, Department of Urology, Minneapolis, Minnesota
  - Division of urology, Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Department of Urology,Vanderbilt University, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - UTHSA - Mays Cancer Center, San Antonio, Texas
- Canada (2):
  - The prostate centre- Diamond Health care centre, Vancouver, British Columbia
  - London Health Sciences Centre Victoria Hospital, London, Ontario

IPD SHARING:
Plan to Share IPD: No